CLINICAL TRIAL: NCT03535610
Title: Uterine Artery Embolization With Microspheres in Patients With Leiomyoma.
Acronym: EMBOSOFT I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Scitech Produtos Medicos Ltda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SC-ES_001
Record Dates: First submitted 2018-05-14; First posted 2018-05-24 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Uterine Leiomyoma
Keywords: Embolization; Uterine Leiomyoma; Embospheres; Microspheres
MeSH Terms: conditions — Myofibroma | interventions — Uterine Artery Embolization

STUDY DESIGN:
Intervention Model Description: Prospective, single-arm, open label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Embolization (Experimental): Uterine Embolization with PVA Microspheres
  Interventions: Device: Uterine Embolization

INTERVENTIONS:
Device: Uterine Embolization — Uterine Embolization with PVA Microspheres

SUMMARY:
To evaluate the therapeutic response to uterine artery embolization in 30 patients with leiomyoma using the microspheres Embosoft (Embosoft® - Scitech Medical).

ELIGIBILITY:
Inclusion Criteria:

* female patients from 18 to 50 years old;
* symptomatic uterine intramural leiomyomas or multiple symptomatic leiomyomas in the presence of intramural;
* patient agrees with study procedures;
* patient signs the informed consent form.

Exclusion Criteria:

* asymptomatic women;
* isolated adenomyosis, pediculated subserous myoma, submucous leiomyoma (50% of uterine cavity diameter), intraligamentous leiomyoma;
* leiomyoma diameter higher than 10 cm;
* leiomyoma above the umbilical scar;
* endometrial neoplasia or hyperplasia or presence of any malignancy
* pregnant or breast feeding women;
* active vasculitis;
* pelvic irradiation history;
* uncontrolled coagulopathies;
* renal insufficiency;
* contrast allergy;
* concomitant use of GnRH analogues.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female patients with Uterine Leiomyoma
Enrollment: 32 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-05-20 (Actual)

PRIMARY OUTCOMES:
Uterine Volume Reduction | 6 months
  Uterine Volume Reduction measured by MRI
Fibroid Reduction | 6 months
  Fibroid Reduction measured by MRI

SECONDARY OUTCOMES:
Quality of Life Improvement | 6 months
  Quality of Life Improvement measured by UFS-QOL
Ovarian Function | 6 months
  Ovarian Function measured by Anti-Mullerian Hormon dosage pre and post-procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Certa Centro de Referência em Tratamentos Avançados, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No